CLINICAL TRIAL: NCT03089359
Title: Prehospital Recognition and Identification of Unspecific Symptoms
Acronym: PRIUS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Katarina Bohm, PhD, Karolinska Institutet
Other Study IDs: PRIUS
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Serious Condition; Morality
Keywords: Unspecific symptoms; Soluvent urokinase plasminogen activator receptor; Lactate; Emergency Medical Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the predictive value of soluvent urokinase plasminogen activator receptor (suPAR) and lactate with respect to serious conditions among patients presenting to the EMS with unspecific symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Unspecific symptoms (not feeling well, decreased general health condition, unable to cope with usual daily activities, feeling weak)
* Normal vital signs
* Transported to ED
* Able to give informed consent/ Next of kin gives informed consent

Exclusion Criteria:

* Specific symptoms
* under 18 years of age
* Stays home / other caregiver than ED
* Referral from caregiver
* No personal numer (social security number)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Unspecific symptoms presenting to the EMS
Sampling Method: Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Serious condition | During medical care event
  Predefined serious condition

SECONDARY OUTCOMES:
Mortality | 24hours and 30 days
  24h and 30 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Bohm, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Helsinki University, Helsinki, Finland
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ivic R, Nurmi J, Kurland L, Vicente V, Lindstrom V, Djarv T, Kaartinen J, Castren M, Bohm K. Soluble urokinase plasminogen activator receptor and lactate as prognostic biomarkers in patients presenting with non-specific chief complaints in the pre-hospital setting - the PRIUS-study. Scand J Trauma Resusc Emerg Med. 2021 Aug 12;29(1):116. doi: 10.1186/s13049-021-00908-z. PMID 34384460